CLINICAL TRIAL: NCT06485271
Title: A Real-world Study of Camrelizumab Alone or in Combination With Apatinib/Chemotherapy for Advanced Gastric Cancer
Status: Recruiting | Type: Observational
Sponsor: Changzhi People's Hospital Affiliated to Changzhi Medical College (Other)
Responsible Party: Sponsor
Other Study IDs: Gastric cancer-RWS
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Gastric Cancer; RWS; PD-1 Immunotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — camrelizumab; apatinib; Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- cohort 1: First-line
  Interventions: Drug: Camrelizumab; Drug: apatinib; Drug: chemotherapy
- cohort 2: Second-line
  Interventions: Drug: Camrelizumab; Drug: apatinib; Drug: chemotherapy
- cohort 3: Third-line and above
  Interventions: Drug: Camrelizumab; Drug: apatinib; Drug: chemotherapy

INTERVENTIONS:
Drug: Camrelizumab — 200mg,iv,d1,Q2W/Q3W
Drug: apatinib — 250mg,qd
Drug: chemotherapy — Standard treatment

SUMMARY:
The purpose of this observational study is to evaluate the safety and efficacy of camrelizumab and apatinib in patients with advanced gastric cancer under real-life conditions, particularly in various subgroups of gastric cancer patients, with a view to providing information about the treatment modalities and efficacy of the treatment in real-life gastric cancer patients and to explore the possible predictive biomarkers of prognosis.Patients, who had both decided to be treated with camrelizumab or apatinib prior to enrollment, were entered into one of the following three cohorts at the discretion of the investigator, based on their disease stage and prior treatment

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, both male and female;
2. patients with advanced gastric cancer diagnosed by pathology or histology and progressed or recurred after 6 months of adjuvant therapy can also be considered for enrollment;
3. Have at least one measurable lesion on imaging (RECIST 1.1 criteria), the spiral CT or MR target lesion should be ≥10 mm and lymph node ≥15 mm;
4. The investigator determines that the patient is amenable to treatment with karelizumab or apatinib;
5. Voluntary enrollment; good compliance and willingness to cooperate with follow-up.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Previous use of other immunotherapy drugs (e.g. PD-1 monoclonal antibody, PD-L1 monoclonal antibody, CTLA4 monoclonal antibody, etc.);
3. Prior use of other anti-angiogenic therapeutic agents (e.g., apatinib, etc.);
4. Patients who, in the judgment of the investigator, are not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced gastric cancer confirmed by pathology or histology
Sampling Method: Probability Sample
Enrollment: 504 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 24 months
  The percentage of subjects achieving complete or partial response in a real-world clinical setting.

SECONDARY OUTCOMES:
Progression free survival | 24 months
  From date of admission until the date of first documented progression in the real-world setting or date of death from any cause, whichever came first, assessed up to 24 months.
Disease control rate | 24 months
  The percentage of subjects achieving complete response, partial response, or disease stability in a real-world clinical setting.
Overall survival | 24 months
  From date of admission until the date of death from any cause, assessed up to 24 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Changzhi People's Hospital Affiliated to Changzhi Medical College, Changzhi, Shanxi, China

IPD SHARING:
Plan to Share IPD: No